CLINICAL TRIAL: NCT00501930
Title: A Randomized, Placebo-Controlled, Double-Blind, Repeat Dose, Dose Escalation Trial to Investigate the Safety, Tolerability and Pharmacokinetics of Supratherapeutic Doses of GSK189075 Administered for 3 Days in Healthy Volunteers
Brief Title: A Study to Evaluate and Study Drug Levels in Blood Plasma When Giving High Doses of GSK189075 to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KG2109799
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes Mellitus, Type 2
Keywords: Dose Escalation;; Supratherapeutic;; GSK189075;; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK189075

SUMMARY:
This study will assess safety and tolerability when taking GSK189075 at doses that are likely to be higher than the expected prescribed doses. The study will also measure the level of GSK189075 in blood after dosing as well as the effect of the drug on certain laboratory tests performed on volunteer urine and blood. Each volunteer will take part in 3 dosing periods and will be given a different dose level at each period (either 2000mg, 4000mg, or a placebo). Volunteers will not know which of the three doses they are receiving. In each period, volunteers will dose every morning for three straight days. Before and after dosing, blood pressure, heart rate, laboratory tests on blood and urine, physical examinations and ECGs will be taken to assess safety. Volunteers will also be asked to provide information should they feel they are having a possible effect from the GSK189075. The levels of GSK189075 in the blood will be assessed by multiple blood draws, most of these will follow the third dose in each period. Depending on the results from the preceding periods, a fourth period may be added to the study to assess another dose level. The fourth period, if this is to occur, will be the same design as the other three periods, and the dose received will be less than 4000mg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and non-pregnant females as determined by a physician on the basis of medical history (including family history of heart disease), physical examination, and clinical laboratory tests.
* written consent given
* agreement to follow specific requirements of birth control during participation.

Exclusion Criteria:

* history of drug or alcohol abuse within one year of the study screening.
* use of tobacco or nicotine-containing products with 6 months prior to the study screening.
* use of any prescription or non-prescription drugs, vitamins, herbal, and dietary supplements within 14 days of the start of the study.
* blood donation within 56 days before the start of the study
* receiving other investigational drugs or participating in other research trials within 30 days of the start of this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-04

PRIMARY OUTCOMES:
Clinical laboratory tests, ECGs, adverse events | screening, Day -1 - 3 all periods, follow up

SECONDARY OUTCOMES:
blood plasma levels of GSK189075 | Day 3
clinical lab tests | each day

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Madison, Wisconsin, United States